Alcon - Business Use Only Protocol - Clinical

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 20-Jul-2018

**Document:** TDOC-0055359  Status: Effective



Title:

# Two Daily Disposable Contact Lenses in Symptomatic Patients

| Protocol Number: | CLS312-P001 / NCT03628599 | |
|---|---|---|
| Sponsor Name and Address: | Alcon Research, Ltd.<br>6201 South Freeway<br>Fort Worth, Texas 76134-2099 | |
| Test Product(s): | DAILIES TOTAL1® Water Gradient silicon hydrodisposable contact lenses (DAILIES TOTAL1) | gel daily |
| Investigator Agreement: | I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Additionally, I will comply with all procedures for data recording and reporting, will permit monitoring, auditing, and inspection of my research center, and will retain all records until notified by the Sponsor. | |
| Principal Investigator: | • | |
| | Signature | Date |
| Name: | | |
| Address: | | |

Printed By: Print Date:

SEE Protocol Template, Vision Care version 2.0, approved 09 SEP 2017

**Document:** TDOC-0055359 **Version:** 1.0; CURRENT; Most-Recent; Effective

Status: Effective 

Effective Date: 20-Jul-2018

# 1 PROTOCOL SYNOPSIS

| Trial Sponsor | Alcon Research, Ltd. |
|---|---|
| | 6201 South Freeway |
| | Fort Worth, Texas 76134-2099 |
| Name of Test Product(s) | DAILIES TOTAL1 Water Gradient silicon hydrogel daily |
| 1 (411) | disposable contact lenses (DAILIES TOTAL1) |
| Name of Control | ACUVUE OASYS® 1-DAY with HydraLuxe™ Technology |
| Product(s) | (Acuvue Oasys 1-Day) |
| Title of Trial | Two Daily Disposable Contact Lenses in Symptomatic |
| | Patients |
| Protocol Number | CLS312-P001 |
| Number of Sites | ~4 |
| Country | US |
| Planned Duration of | Test Product: 28 days (±2 days) |
| Exposure | Control Product: 28 days (±2 days) |
| Number of Subjects | Target to complete: 30 |
| | Planned to enroll: ~36 |
| Study Population | Volunteer subjects aged 18 or over who are symptomatic |
| | contact lens wearers and who wear their habitual monthly or |
| | bi-weekly replacement lenses at least 3 days per week and at |
| | least 5 hours per day |
| Objective(s) | The overall objective of the study is to evaluate the |
| | performance of Acuvue Oasys 1-Day and DAILIES |
| | TOTAL1 with respect to visual acuity, |
| | in a symptomatic study population of monthly or |
| | bi-weekly replacement lens wearers |
| Endpoints | Primary Effectiveness |
| | • VA (4-Week Follow-up) |

Effective Date: 20-Jul-2018 Version: 1.0; CURRENT; Most-Recent; Effective

**Document:** TDOC-0055359  Status: Effective

| | Safety | |
|---|---|---|
| | AEs Diamigrassany findings | |
| | <ul><li>Biomicroscopy findings</li><li>Device deficiencies</li></ul> | |
| Assessments | Effectiveness | |
| | • VA (Snellen distance) | |
| | Manifest refraction | _ |
| | BCVA (Snellen distance) | e with manifest refraction) |
| | Safety • AEs | |
| | <ul><li>AEs</li><li>Biomicroscopy</li></ul> | |
| | <ul><li>Device deficiencies</li></ul> | |
| Study Design | Prospective | Single-masked |
| , <u>,</u> | Single group | (trial subject) |
| | Parallel group | Single-masked |
| | Crossover | (Investigator) |
| | Other | Double-masked |

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 20-Jul-2018

**Document:** TDOC-0055359  Status: Effective

| | | Open-label |
|---|---|---|
| | | Other |
| | ☐ Contralateral | Randomized |
| | ⊠ Bilateral | |
| | ☐ Monocular lens wear | |
| Test Product Details | Primary | delefilcon A |
| | component/material | |
| | Product Name | DAILIES TOTAL1 |
| | Manufacturer | Alcon |
| | Other | The lenses will be available in -2.00 D to -6.00 D in 0.25 D steps and -6.50 D to -8.50 D in 0.50 D steps |
| Control Product Details | Primary | senofilcon A |
| | component/material | |
| | Product Name | Acuvue Oasys 1-Day |
| | Manufacturer | Johnson & Johnson |
| | Other | The lenses will be available in -2.00 D to -6.00 D in 0.25 D steps and -6.50 D to -8.50 D in 0.50 D steps |
| Inclusion Criteria | 1. Subject must be at least | t 18 years of age. |
| | 2. Subject must be able to | understand and must sign an ICF |
| | that has been approved | by an IRB. |
| | 4 Soft contact lens weare | rs in both eyes during the past 3 |
| | months. | is in both eyes during the past 5 |
| | <ul><li>5. Manifest cylinder ≤ 0.7</li></ul> | '5 D in each eve. |
| | 6. BCVA 20/25 or better | • |
| | | g to wear the study lenses at least |
| | 3 days per week and at | • |
| | 8. Subject must be willing to stop wearing their had contact lenses for the duration of study participation. | |
| Exclusion Criteria | Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator. | |


Status: Effective 

| | drops will be permitted as needed but not provided. |
|---|---|
| Associated Materials | No lens care products will be used. Commercial re-wetting |
| | vision). |
| | 14. Monocular subjects (only one eye with functional |
| | previous 30 days or currently enrolled in any clinical trial. |
| | 13. Participation of the subject in a clinical trial within the |
| | aforementioned persons may not participate in the study. |
| | or individuals living in the households of the |
| | Investigator, family members of the Investigator's staff, |
| | 12. The Investigator, his/her staff, family members of the |
| | instillation during contact lens wear. |
| | 11. Any use of topical ocular medications that would require |
| | per week) over the last 3 months prior to enrollment. |
| | modality (routinely sleeping in lenses for at least 1 night |
| | 10. Wearing habitual contact lenses in an extended wear |
| | 9. Current or history of intolerance, hypersensitivity, or allergy to any component of the study products. |
| | prior to enrollment for this trial. Of Current or history of intelerance hypergeneitivity, or |
| | 8. Eye injury in either eye within 12 weeks immediately |
| | 7. Current or history of herpetic keratitis in either eye. |
| | contact lens wear. |
| | that, in the opinion of the Investigator, would preclude |
| | 6. Current or history of pathologically dry eye in either eye |
| | mild (Grade 2) or higher. |
| | (Grade 3) or higher and/or corneal vascularization that is |
| | 5. Biomicroscopy findings at screening that are moderate |
| | during the study. |
| | punctal plugs) within the previous 12 months or planned |
| | 4. Ocular or intraocular surgery (excluding placement of |
| | surgery during the study or irregular cornea in either eye. |
| | 3. History of refractive surgery or plan to have refractive |
| | contact lens wear could be contraindicated, as determined by the Investigator. |
| | contest long wear could be controlled as |

Alcon - Business Use Only Protocol - Clinical


Status: Effective 

Effective Date: 20-Jul-2018

 Table 1-1
 Schedule of Study Procedures and Assessments

| Procedure/ Assessment | | Visit 1<br>(Day 1) | Visit 2 (Day 7 ± 2 days) | Visit 3 (Day 28 ± 2 days) | led Visit | Exit |
|---|---|---|---|---|---|---|
| | Pre-screening | Baseline /<br>Fitting /<br>Dispense | 1-week<br>Follow-up | 4-week<br>Follow-up<br>/ Exit | Unscheduled Visit | Early Exit |
| Informed Consent | - | ✓ | - | - | - | - |
| Demographics | - | ✓ | - | - | - | - |
| Medical History | - | ✓ | ✓ | ✓ | <b>✓</b> | ✓ |
| Concomitant Medications | - | ✓ | (✓) | <b>(</b> ✓) | <b>(√)</b> | <b>(√)</b> |
| Inclusion/Exclusion | - | ✓ | - | - | - | - |
| VA w/ habitual correction (OD, OS, Snellen distance)* | - | √a | - | - | - | - |
| Manifest refraction* | - | ✓ | (✓) | <b>(</b> ✓) | <b>(√)</b> | <b>(√)</b> |
| BCVA (OD, OS, Snellen distance with manifest refraction)* | - | <b>√</b> | <b>(</b> ✓) | ( <b>v</b> ) | <b>(</b> ✓) | <b>(✓)</b> |
| Biomicroscopy | - | ✓ | ✓ | ✓ | ✓ | ✓ |
| Dispense study lenses | - | ✓ | - | - | ı | - |
| VA w/ study lenses (OD, OS, Snellen distance) | - | ✓ | ✓ | ✓ | <b>(✓)</b> | ✓ |

Alcon - Business Use Only Protocol - Clinical


Status: Effective 

Effective Date: 20-Jul-2018

| Procedure/ Assessment | eening | Visit 1<br>(Day 1) | Visit 2 (Day 7 ± 2 days) | Visit 3 (Day 28 ± 2 days) | lled Visit | Exit |
|---|---|---|---|---|---|---|
| | Pre-screening | Baseline /<br>Fitting /<br>Dispense | 1-week<br>Follow-up | 4-week<br>Follow-up<br>/ Exit | Unscheduled | Early Exit |
| AEs | - | ✓ | ✓ | ✓ | ✓ | ✓ |
| Device deficiencies | - | ✓ | ✓ | ✓ | ✓ | ✓ |
| Exit Form | - | <b>(✓)</b> | <b>(√)</b> | <b>(√)</b> | <b>(√)</b> | ✓ |

<sup>&</sup>lt;sup>a</sup> Performed based on habitual lenses

<sup>(✓)</sup> assessment performed as necessary, eg, decrease of VA by 2 lines or more with investigational product (IP)

<sup>\*</sup> Source only


Status: Effective 

# 1.1 Abbreviations

| Abbreviation | Definition |
|---|---|
| Acuvue Oasys | ACUVUE OASYS 1-DAY with HydraLuxe Technology |
| 1-Day or | |
| AO1D | |
| ADE | Adverse device effect |
| AE | Adverse event |
| ASADE | Anticipated serious adverse device effect |
| BCVA | Best corrected visual acuity |
| CFR | Code of Federal Regulations |
| CL | Contact lens |
| D | Diopter |
| D/C | Discontinue |
| DAILIES | DAILIES TOTAL1 Water Gradient silicon hydrogel daily disposable |
| TOTAL1 or | contact lenses |
| DT1 | |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| LogMAR | Logarithm of the minimum angle of resolution |
| mm | Millimeter |
| MOP | Manual of procedures |
| N/A | Not applicable |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |
| SAE | Serious adverse event |
| SADE | Serious adverse device effect |
| US | United States |
| USADE | Unanticipated serious adverse device effect |
| VA | Visual acuity |

Effective Date: 20-Jul-2018


**Document:** TDOC-0055359

Status: Effective

2 TABLE OF CONTENTS

| Tw | o Daily I | Disposable Contact Lenses in Symptomatic Patients | 1 |
|---|---|---|---|
| 1 | PROTO | COL SYNOPSIS | 2 |
| | 1.1 | Abbreviations | 8 |
| 2 | TABLE | OF CONTENTS | 9 |
| Lis | t of Table | es | 11 |
| Lis | t of Figu | res | 11 |
| 3 | INTROI | DUCTION | 12 |
| | 3.1 | Study Rationale and Purpose | 12 |
| | 3.2 | Trial Objective | |
| | 3.3 | Risks and Benefits | |
| | 3.4 | Subject Population | 13 |
| | 3.5 | Outline of Study | |
| 4 | TREAT | MENTS ADMINISTERED | 14 |
| | 4.1 | Identity of Study Treatments | 14 |
| | 4.2 | Accountability Procedures | 15 |
| 5 | STUDY | PROCEDURES AND ASSESSMENTS | 16 |
| | 5.1 | Visits and Examinations | 16 |
| | | 5.1.1 Visit 1 (Day 1) – Baseline/Fitting/Dispense | 16 |
| | | 5.1.2 Visit 2 (Day $7 \pm 2$ Days) – 1-Week Follow-up | 18 |
| | | 5.1.3 Visit 3 (Day $28 \pm 2$ Days) $-4$ -Week Follow-up / Exit | 20 |
| | 5.2 | Unscheduled Visits | 21 |
| | 5.3 | Discontinued Subjects | 22 |
| | 5.4 | Clinical Study Termination | 22 |
| 6 | ANALY | SIS PLAN | 23 |
| | 6.1 | Subject Evaluability | 23 |
| | 6.2 | Analysis Data Sets | 23 |
| | | 6.2.1 Safety Analysis Set | 23 |
| | 6.3 | Demographic and Baseline Characteristics | 24 |
| | 6.4 | Effectiveness Analyses | 24 |
| | | 6.4.1 Primary Effectiveness | 24 |
| | | 6.4.1.1 Statistical Hypotheses | 24 |

Alcon - Business Use Only Protocol - Clinical

Effective Date: 20-Jul-2018


| Sta | tus: Effective | e | |
|---|---|---|---|
| | | 6.4.1.2 Analysis Methods | 24 |
| | | | 24 |
| | | | 25 |
| | 6.5 | Subgroup Analyses | 25 |
| | 6.6 | Handling of Missing Data | |
| | 6.7 | Multiplicity | |
| | 6.8 | Safety Analysis | |
| | 6.9 | Interim Analyses | |
| | 6.10 | Sample Size Justification. | |
| 7 | | SE EVENTS AND DEVICE DEFICIENCIES | |
| • | 7.1 | General Information | |
| | 7.1 | Monitoring for Adverse Events | |
| | 7.2 | Procedures for Recording and Reporting | |
| | 7.4 | Return product analysis | |
| | 7.5 | Follow-Up of Subjects with Adverse Events | |
| | 7.6 | Pregnancy in the Clinical Study | |
| 8 | | DENTIALITY, BIAS, AND MASKING | |
| O | 8.1 | Subject Confidentiality and Methods Used to Minimize Bias | |
| | 8.2 | Unmasking of the Study Treatment | |
| 9 | | ANDLING AND ADMINISTRATIVE REQUIREMENTS | |
| 7 | | | |
| | 9.1 | Completion of Source Documents and Case Report Forms | |
| | 9.2 | Data Review and Clarifications | |
| 10 | 9.3 | Regulatory Documentation and Records Retention | |
| 10 | | AND COMPLIANCE | |
| | 10.1 | Compliance | |
| | 10.2 | Institutional Review Board (IRB) | |
| 11 | PROTO | COL AMENDMENT HISTORY | 39 |
| 12 | REFERE | ENCES | 39 |
| | 12.1 | References applicable for all clinical trials | 39 |
| | | 12.1.1 US references applicable for clinical trials | 39 |
| | 12.2 | References for this clinical trial | 39 |

| T11 11 | List of Tables | ( |
|------------|----------------------------------------------|----|
| Table 1-1 | Schedule of Study Procedures and Assessments | 0 |
| | List of Figures | |
| Figure 7–1 | Categorization of All AEs | 29 |
| Figure 7-2 | Categorization of All Serious Adverse Events | 30 |

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 20-Jul-2018


Alcon - Business Use Only Protocol - Clinical

**Document:** TDOC-0055359

Status: Effective


Status: Effective 

#### 3 INTRODUCTION

### 3.1 Study Rationale and Purpose

The contact lenses for this study are intended for the optical correction of refractive myopia in persons with non-diseased eyes who are dryness symptomatic with their habitual weekly/monthly contact lenses.

The primary purpose of this study is to conduct a pilot study with DAILIES TOTAL1 and Acuvue Oasys 1-Day to guide the protocol development of the subsequent larger scale head-to-head phase 4 trial. Additionally, this study is being conducted to re-fit habitual weekly/monthly symptomatic wearers into DAILIES TOTAL1 and Acuvue Oasys 1-Day

The primary endpoint was selected to support the overall study objective. Procedures for measurement of this endpoint are standard in eye care professional practice. The design of this study is justified based upon preclinical and clinical testing, as described within the product's Instructions for Use. Acuvue Oasys 1-Day contact lenses were chosen as the control product because these lenses have the same wear modality and a similar material to the DAILIES TOTAL1 lenses.

There are no immediate plans to submit the results of this study for publication; however, the results may be offered for publication if they are of scientific interest, or if the results relate to a product that is subsequently approved or cleared for marketing.

# 3.2 Trial Objective

| The overall objective of the study is to evaluate the performance | of DAILIES TOTAL1 and |
|---|---|
| Acuvue Oasys 1-Day with respect to VA, | in a symptomatic study |
| population of monthly or bi-weekly replacement lens wearers. | |

The primary objective is to evaluate VA after approximately 4 weeks of lens wear.



Data collected may be used for the sample size calculation of a claims trial with DAILIES TOTAL1 and Acuvue Oasys 1-Day.


Status: Effective 

The safety objective is to describe the safety profile of the investigational products through evaluation of AEs, biomicroscopy findings, and device deficiencies.

#### 3.3 Risks and Benefits

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. There is no intended clinical benefit to the subject; additionally, both study lenses have the potential to reduce dryness symptoms while wearing contact lenses. Material properties and design characteristics of the contact lens in development are features consistent with successful contact lens wear.

DAILIES TOTAL1 and ACUVUE OASYS 1-DAY contact lenses are for daily wear use under a daily disposable wear modality; further details on any known potential risks and benefits can be found in the package inserts.

The DAILIES TOTAL1 and Acuvue Oasys 1-Day contact lenses are not intended for use with a cleaning/disinfecting solution, and the biocompatibility with lens care solutions and any associated clinical effects are unknown.

A summary of the known potential risks and benefits associated with DAILIES TOTAL1 lenses can be found in the package insert. Risks are minimized by compliance with the eligibility criteria and study procedures, and through close supervision by a licensed clinician during exposure to the study lenses. The potential harms associated with on-eye exposure to the new lens materials include toxicity response, blurred vision, and ocular discomfort. In general, the risks with the contact lens are anticipated to be similar to other marketed daily disposable soft contact lenses.

The site personnel will educate subjects on proper hygiene and lens handling, and compliance with the use of contact lenses according to the protocol. Subjects should be instructed not to wear contact lenses while sleeping or swimming. The site personnel will also advise the subjects to remove contact lenses and return for prompt follow-up of symptoms, such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.

# 3.4 Subject Population

The study population includes approximately 36 volunteer subjects to be enrolled at approximately 4 sites, with approximately 9 subjects enrolled per site. The study population will consist of subjects aged 18 or over with normal eyes (other than the need for optical correction for myopia), who are adapted, existing wearers of weekly/monthly soft contact lenses in both eyes and positive for dryness symptoms with their habitual contact lenses


Status: Effective 

Subjects may be pre-screened for dryness symptoms and must be screened according to the full list of inclusion/exclusion criteria in Section 1 of this protocol. Rescreening of subjects is not allowed in this study.

### 3.5 Outline of Study

This will be a prospective, multi-site, randomized, parallel-group, open-label study comparing 2 daily disposable contact lenses. The expected duration of subject participation in the study is approximately 4 weeks, with 3 scheduled visits. The study is expected to be completed in approximately 8 weeks.

#### 4 TREATMENTS ADMINISTERED

Subjects will be randomized in a 1:1 manner to receive treatment with DAILIES TOTAL1 or Acuvue Oasys 1-Day.

# 4.1 Identity of Study Treatments

| DESCRIPTION OF TEST AND CONTROL PRODUCTS | | |
|---|---|---|
| | Test Lens | Control Lens |
| Lens | DAILIES TOTAL1 | Acuvue Oasys 1-Day |
| Material | delefilcon A | senofilcon A |
| Water Content | 33% | 38% |
| Base Curve (mm) | 8.5 | 8.5 and 9.0 |
| Diameter (mm) | 14.1 | 14.3 |
| Rx powers to be available in this study | -2.00 D to -6.00 D in<br>0.25 D steps and -6.50 D<br>to -8.50 D in 0.50 D steps | -2.00 D to -6.00 D in<br>0.25 D steps and -6.50 D<br>to -8.50 D in 0.50 D steps |
| Packaging, Labeling, and Supply | <ul> <li>Blister foil pack</li> <li>Commercial foil</li> <li>Commercial Packaging</li> <li>Lenses will be provided in 30 count boxes per power.</li> <li>Lenses should be stored at room temperature.</li> </ul> | <ul> <li>Blister foil pack</li> <li>Commercial foil</li> <li>Commercial Packaging</li> <li>Sites will procure the control lenses.</li> <li>Lenses should be stored at room temperature.</li> </ul> |


Status: Effective 

| Usage | • | Wear: |
|-------|---|-------------------------------------------------------------|
| | | <ul> <li>Daily wear</li> </ul> |
| | | <ul> <li>Bilateral, parallel group</li> </ul> |
| | • | Replacement period: daily disposable |
| | • | Exposure: Goal is at least 8 hours per day, at least 3 days |
| | | per week over a 4-week period |
| | • | Lens Care: N/A |

### 4.2 Accountability Procedures

Upon receipt of the study lenses, the Investigator or delegate will conduct an inventory. Designated study staff will provide the study lenses to the subjects in accordance with their randomization schedule. Throughout the study, the Investigator or delegate must maintain records of study treatment dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of clinical supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation.

It is the Investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All used foils and unused supplies are returned by each subject
- All unused products are available for return to the Study Sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related adverse event [ie, ADE or SADE] are returned to the Study Sponsor for investigation. Refer to Section 7.3 of this protocol for additional information on the reporting of device deficiencies and AEs and the return of study products associated with these events.


Status: Effective 

Effective Date: 20-Jul-2018

#### 5 STUDY PROCEDURES AND ASSESSMENTS

#### 5.1 Visits and Examinations

# 5.1.1 Visit 1 (Day 1) – Baseline/Fitting/Dispense



Obtain demographic information and medical history, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications.

- 5 Perform Snellen VA with habitual correction (in source).
  - OD, OS, distance only, contact lenses
  - Over-refraction if necessary to determine the best contact lens-corrected VA and determine final study lens power(s)
- 6 Perform a manifest refraction (in source)
- 7 Perform Snellen BCVA with manifest refraction (in source).
  - OD, OS, distance only

Note: Distance BCVA must be 20/25 or better in each eye for the subject to qualify for the study.

Alcon - Business Use Only Protocol - Clinical


Status: Effective 

Effective Date: 20-Jul-2018

Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: Limbal hyperemia Bulbar hyperemia Corneal staining Conjunctival staining Palpebral conjunctival observations Corneal epithelial edema Corneal stromal edema Corneal vascularization Conjunctival compression/indention Chemosis Corneal infiltrates Other findings 9 Determine study lens powers based upon the manifest refraction and habitual lens powers. 10 Review inclusion/exclusion criteria to determine if the subject qualifies to be randomized into the study. If subject qualifies, request randomization. If subject does not qualify, exit the subject from the study as a screen failure. 11 Based upon the randomized treatment assignment, have the subject insert the appropriate study lenses. Keep all lidding foils of lenses used during lens fit process for study lens accountability. Evaluate the study lenses by performing the following: 12 Snellen VA with study lenses (OD and OS, at distance)\* \*VA w/study lenses must be 20/40 OU or better for subject to leave the office 15 Assess and record any AEs and device deficiencies reported or observed during the study visit.


Status: Effective 

| | Note: AEs and device deficiencies must be recorded for all enrolled subjects from the time of signature of informed consent including those that screen fail. |
|---|---|
| 16 | Dispense study lenses. Provide the subject with written and verbal instructions on |
| | lens wear. |
| | Verbal instruction only: If the subject experience an unusual feeling after lens |
| | insertion (ie, discomfort), the lens may be inverted. Remove and insert the lens |
| | again. |
| 17 | Schedule Visit 2 to take place after $7 \pm 2$ days of lens wear. |
| 18 | Note: If for some reason a subject is unable to wear a study lens for the duration of this visit |
| | window, instruct the subject to return to the site for an Unscheduled Visit, including, if |
| | possible, lens removal on site. The subject should then be scheduled to return to the clinic |
| | for Visit 2 (if possible) or exited from the study. |

# 5.1.2 Visit 2 (Day $7 \pm 2$ Days) – 1-Week Follow-up

| 1 | Obtain information on any changes in medical health and/or the use of concomitant |
|---|---|
| | medications. |
| 2 | Record any device deficiencies or AEs, including those associated with changes in |
| | concomitant medication dosing, which are observed or reported since the previous |
| | visit. |
| 3 | Review subject compliance with lens wear and adjunct product usage. |
| 3 | Review subject compliance with tens wear and adjunct product usage. |
| 5 | Perform a manifest refraction (as needed) (in source) |
| 6 | Perform Snellen BCVA with manifest refraction (as needed) (in source) |
| | OD, OS, distance only |
| | Note: Perform BCVA if there is a decrease of VA by 2 lines or more with IP |
| 7 | Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: |
| | Limbal hyperemia |
| | Bulbar hyperemia |
| | Corneal staining |
| | Conjunctival staining |
| | Palpebral conjunctival observations |
| | Corneal epithelial edema |
| | Corneal stromal edema |
| | Corneal vascularization |

Alcon - Business Use Only Protocol - Clinical


Status: Effective 

Effective Date: 20-Jul-2018

Conjunctival compression/indention Chemosis Corneal infiltrates Other findings Evaluate the study lenses by performing the following: 8 • Snellen VA with study lenses (OD and OS, at distance) 12 Assess and record any AEs and device deficiencies reported or observed during the study visit. Note: AEs and device deficiencies must be recorded for all enrolled subjects from the time of signature of informed consent regardless of their enrollment status (screen failure or randomized). 13 Schedule Visit 3 to take place after 28± 2 days of lens wear 14 Note: If for some reason a subject is unable to wear a study lens for the duration of this visit window, instruct the subject to return to the site for an Unscheduled Visit, including, if possible, lens removal on site. The subject should then be scheduled to return to the clinic

Printed By: Print Date:

for Visit 3 (if possible) or exited from the study.


Status: Effective 

Effective Date: 20-Jul-2018

# 5.1.3 Visit 3 (Day $28 \pm 2$ Days) – 4-Week Follow-up / Exit

| 1 | Obtain information on any changes in medical health and/or the use of concomitant |
|---|---|
| | medications. |
| 2 | Record any device deficiencies or AEs, including those associated with changes in |
| | concomitant medication dosing, which are observed or reported since the previous |
| | visit(s). |
| 3 | Review subject compliance with lens wear and adjunct product usage. |
| 5 | Perform a manifest refraction (as needed) (in source) |
| 6 | Perform Snellen BCVA with manifest refraction (as needed) (in source) |
| | • OD, OS, distance only |
| | Note: Perform BCVA if there is a decrease of VA by 2 lines or more with IP |
| 7 | Perform slit-lamp biomicroscopy (without contact lenses) to evaluate the following: |
| | Limbal hyperemia |
| | Bulbar hyperemia |
| | Corneal staining |
| | Conjunctival staining |
| | Palpebral conjunctival observations |
| | Corneal epithelial edema |
| | Corneal stromal edema |
| | Corneal vascularization |
| | Conjunctival compression/indention |
| | • Chemosis |
| | Corneal infiltrates |
| | • Other findings |
| 8 | Evaluate the study lenses by performing the following: |
| | • Snellen VA with study lenses (OD and OS, at distance) |


Status: Effective 

Effective Date: 20-Jul-2018



#### 5.2 Unscheduled Visits

Any visit that occurs between regularly scheduled visits is an Unscheduled Visit. If a subject requires an Unscheduled Visit, he/she must be advised to return to the office wearing the study lenses, if at all possible (unless he/she is experiencing a sign or symptom [as indicated in Section 3.3 Risks and Benefits]). During all unscheduled visits, the Investigator must conduct the following procedures:

- Collect AE and device deficiency information
- Assess and record changes in medical condition or concomitant medication
- Assess and record VAs


Status: Effective 

Perform biomicroscopy (assessments with or without lenses, as possible)

In addition, all procedures for Visit 3 (4-Week Follow-up/Exit) should be completed (as possible). The Investigator may perform additional procedures for proper diagnosis and treatment of the subject. The Investigator must document this information in the subject's case history source documents.

If during an Unscheduled Visit the subject is discontinuing the study lenses or discontinuing from the study, the Investigator must conduct Exit procedures according to Table 1-1: Schedule of Study Procedures and Assessments, as possible.

### 5.3 Discontinued Subjects

Discontinued subjects are those who withdraw or are withdrawn from the study after signing the informed consent, including screen failures. Subjects may discontinue from the study at any time for any reason. Subjects may also be discontinued from the study at any time if, in the opinion of the Investigator, their continued participation poses a risk to their health. Discontinued subjects will not be replaced (ie, their subject numbers will not be re-assigned/re-used).

Should a subject exhibit any clinically relevant signs, symptoms, or other clinical observations that possibly could be associated with suspected sensitivity or intolerance to one of the study treatments, the Investigator must document those observations on an AE Form.

Any subject who exits early from the study (excluding screen failures) must undergo all procedures outlined at Visit 3, as applicable.

The Investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, Investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 5.4 Clinical Study Termination

The Study Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time, for reasonable cause.


Status: Effective 

If the clinical study is prematurely terminated or suspended by the Study Sponsor:

The Study Sponsor must:

- Immediately notify the Investigator(s) and subsequently provide instructions for study termination.
- Inform the Investigator(s) and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension, as applicable.
- The Investigator must:
  - Promptly notify the IRB of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for post-study treatment options as needed.

The Investigator may terminate a site's participation in the study for reasonable cause.

#### 6 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized with counts and percentages from each category. Any deviations to this analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

# 6.1 Subject Evaluability

The final subject evaluability will be determined prior locking the database, based on the Deviations and Evaluability Plan.

# 6.2 Analysis Data Sets

# **6.2.1** Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed.


Status: Effective 

### 6.3 Demographic and Baseline Characteristics



#### **6.4** Effectiveness Analyses



# 6.4.1 Primary Effectiveness

The primary objective of this study is to evaluate VA after approximately 4 weeks of lens wear. The primary endpoint is distance VA with study lenses, collected in Snellen at the 4-week follow-up visit, for each eye. Conversion will be made to the logMAR scale.

### **6.4.1.1** Statistical Hypotheses

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.

### 6.4.1.2 Analysis Methods

Counts and percentage in each Snellen VA category will be provided, and descriptive statistics (number of observations, mean, standard deviation, median, minimum, maximum) for the logMAR converted values will be presented.




Status: Effective 

Effective Date: 20-Jul-2018



### 6.5 Subgroup Analyses

It is not expected that demographic or baseline characteristics will have an impact on the study results in this study. No subgroup analyses are planned.

# 6.6 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analyses. No imputation for missing values will be carried out.

# 6.7 Multiplicity

No multiplicity adjustment needs to be considered for the effectiveness endpoints since no formal hypothesis testing will be conducted.

# 6.8 Safety Analysis

The safety endpoints for this study are AEs, biomicroscopy findings, and device deficiencies.

Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to


Status: Effective 

study discontinuation, significant non-serious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to study lenses.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (Visit 1) to any subsequent visit will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits for these eyes experiencing the increase.

Two listings (prior to exposure of study lenses and treatment-emergent) of device deficiencies, as recorded on the Device Deficiency Form, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be done for safety analysis.

### 6.9 Interim Analyses

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

# **6.10** Sample Size Justification

For VA with a sample size of 15 in each treatment group, a two-sided 95% confidence interval for the difference of 2 means will extend 0.05 from the observed difference in means with an assumed common standard deviation of 0.07.

Effective Date: 20-Jul-2018 Version: 1.0; CURRENT; Most-Recent; Effective **Document:** TDOC-0055359

 Status: Effective

## 7 ADVERSE EVENTS AND DEVICE DEFICIENCIES

### **Terms and Definitions**

| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or injury, or |
|---|---|
| | untoward clinical signs (including abnormal laboratory findings) in |
| | subjects, users or other persons, whether or not related to the |
| | investigational medical device (test product). Note: For subjects, |
| | this definition includes events related to the test product, the |
| | control product, or the procedures involved. For users or other |
| | persons, this definition is restricted to events related to the test |
| | product. |
| Adverse Device | AE related to the use of an investigational medical device (test |
| Effect (ADE) | product) or control product. Note: This definition includes AEs |
| | resulting from insufficient or inadequate instructions for use, |
| | deployment, implantation, installation, or operation; any |
| | malfunction; and use error or intentional misuse of the test product |
| | or control product. |
| Anticipated Serious | Serious ADE which by its nature, incidence, severity or outcome |
| Adverse Device | has been identified in the risk management file. |
| Effect (ASADE) | |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, |
| | durability, reliability, safety, or performance. Note: This definition |
| | includes malfunctions, use errors, and inadequate labeling. |
| Malfunction | Failure of a medical device to meet its performance specifications |
| | or otherwise perform as intended. Performance specifications |
| | include all claims made in the labeling of the device. The intended |
| | performance of the device refers to the intended use for which the |
| | device is labeled or marketed. |
| Non-serious Adverse | AE that does not meet the criteria for an SAE. |
| Event | |
| Serious Adverse | AE that led to any of the following: |
| Event (SAE) | • Death. |
| | A serious deterioration in the health of the subject that either |
| | resulted in: |
| | a) a life-threatening illness or injury. |
| | Note: Life-threatening means that the individual was at |
| | immediate risk of death from the event as it occurred, ie, it |

Effective Date: 20-Jul-2018 Version: 1.0; CURRENT; Most-Recent; Effective

**Document:** TDOC-0055359  Status: Effective

| | does not include an event which hypothetically might have |
|---|---|
| | caused death had it occurred in a more severe form. |
| | b) any potentially sight-threatening event or permanent |
| | impairment to a body structure or a body function. |
| | c) in-patient hospitalization or prolonged hospitalization. |
| | Note: Planned hospitalization for a pre-existing condition, |
| | without serious deterioration in health, is not considered |
| | an SAE. In general, hospitalization signifies that the |
| | individual remained at the hospital or emergency ward for |
| | observation and/or treatment (usually involving an |
| | overnight stay) that would not have been appropriate in the |
| | physician's office or an out-patient setting. Complications |
| | that occur during hospitalization are adverse events. If a |
| | complication prolongs hospitalization or fulfills any other |
| | serious criteria, the event is serious. When in doubt as to |
| | whether "hospitalization" occurred, the event should be |
| | considered serious. |
| | d) a medical or surgical intervention to prevent a) or b). |
| | e) any indirect harm as a consequence of incorrect diagnostic |
| | test results when used within manufacturer's instructions |
| | for use. |
| | • Fetal distress, fetal death, or a congenital abnormality or birth |
| | defect. |
| | Refer to Section 7.1 for additional SAEs. |
| Serious Adverse | ADE that has resulted in any of the consequences characteristic of |
| Device Effect | an SAE. |
| (SADE) | |
| Significant Non- | A significant non-serious AE is a symptomatic, device-related, |
| Serious Adverse | non-sight threatening AE that warrants discontinuation of any |
| Event | contact lens wear for greater than or equal to 2 weeks. |
| | Refer to Section 7.1 for additional Significant Non-Serious AEs. |
| Unanticipated | Serious adverse device effect which by its nature, incidence, |
| Serious Adverse | severity or outcome has not been identified in the risk management |
| Device Effect | file. |
| (USADE) | |


Status: Effective 

Effective Date: 20-Jul-2018

| Use Error | Act or omission of an act that results in a different medical device |
|---|---|
| | response than intended by manufacturer or expected by user. |
| | Note: This definition includes slips, lapses, and mistakes. An |
| | unexpected physiological response of the subject does not in itself |
| | constitute a use error. |

### 7.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test *product*).

Figure 7–1 Categorization of All AEs



Effective Date: 20-Jul-2018 Document: TDOC-0055359 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective 

Figure 7-2 **Categorization of All Serious Adverse Events** 



#### **Specific Events Relevant to this Protocol**

#### Serious Adverse Events

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the Investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics:
  - Central or paracentral location
  - Penetration of Bowman's membrane
  - Infiltrates > 2 mm diameter
  - **Iritis**
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon


Status: Effective 

- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA [VA w/ study lenses (OD, OS), Snellen distance] from enrollment visit that fails to resolve; this loss should be confirmed with Manifest Refraction BCVA
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

#### Significant Non-Serious Adverse Events

A significant non-serious AE is a symptomatic, device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. In addition, the Investigator must report any occurrence of the following as a Significant Non-Serious AE:

- Peripheral non-progressive non-infectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score greater than or equal to Grade 3
- Temporary vision loss as defined by loss of 2 or more lines of BCVA [VA w/ study lenses (OD, OS), Snellen distance]from enrollment visit that persists for 2 or more weeks this loss should be confirmed with Manifest Refraction BCVA
- Neovascularization score greater than or equal to Grade 2

The above events are based upon the categories provided in the ISO 11980 and the US FDA Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses and Contact Lens Care Products.


Status: Effective 

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with patient harm (ie, ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The Investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any patient harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (eg, incorrect lens power/diameter/base curve/color)
- Lens/solution cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (eg, mislabeled product, tampered seal, leaking bottle/container)
- Suspect product contamination
- Lack of performance

### 7.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking the standard questions:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

Additionally, changes in *any protocol-specific parameters and/or questionnaires* evaluated during the study are to be reviewed by the Investigator. Any untoward (unfavorable and unintended) change in *a protocol-specific parameter or questionnaire response* that is clinically relevant, in the opinion of the Investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

# 7.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any pre-existing medical conditions or signs/symptoms present in a subject prior to the start of the study (ie, before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.


Status: Effective 

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the Investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

- ADEs or SAEs are documented on the Serious Adverse Event and Adverse Device Effect eCRF within 24 hours of the Investigator's or site's awareness.
- Device deficiencies are documented on the Device Deficiency eCRF within 24 hours of the Investigator's or site's awareness.
- A printed copy of the completed *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
- Certificate of Death, etc, if applicable, in narrative section of the *Serious Adverse Event* and *Adverse Device Effect* eCRF.

*Note:* Should the EDC system become non-operational, the site must complete the appropriate paper *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* Form. The completed form is emailed to the Study Sponsor at msus.safety@alcon.com according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

Study Sponsor representatives may be contacted for any protocol related question.

Further, depending upon the nature of the AE or device deficiency being reported, the Study Sponsor may request copies of applicable portions of the subject's medical records. The Investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.


Status: Effective 

#### **Intensity and Causality Assessments**

Where appropriate, the Investigator must assess the intensity (severity) of the AE based upon medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the Investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by Study Sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (ie, there are other more likely causes for the AE).

The Study Sponsor will assess the AEs and may upgrade the Investigator's assessment of seriousness and/or causality. The Study Sponsor will notify the Investigator of any AEs that are upgraded from non-serious to serious or from unrelated to related.

# 7.4 Return product analysis

Alcon products associated with device deficiencies and/or product related AEs should be returned and must include the Complaint # which will be provided by Study Sponsor after the case is entered in the Study Sponsor's Global Product Complaint Management System. These products should be returned to the Sponsor at the end of the study, unless instructed otherwise by the Sponsor.


Status: Effective 

### 7.5 Follow-Up of Subjects with Adverse Events

The Investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The Investigator should provide the Study Sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (ie, database lock).

Any additional data received up to 1 month after subject discontinuation or exit must be documented and available upon the Study Sponsor's request. All complaints received after this time period will be considered and processed as spontaneous and should be communicated to the medical device's manufacturer as per local requirements.

The Investigator should also report complaints on non-Alcon products (ie, the control lenses) directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

## 7.6 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case—by-case basis.

## 8 CONFIDENTIALITY, BIAS, AND MASKING

# 8.1 Subject Confidentiality and Methods Used to Minimize Bias

The Investigator must ensure that the subject's anonymity is maintained throughout the course of the study. In particular, the Investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. At the end of the clinical study, the Sponsor will collect a copy of the enrollment log without any identifying subject information. All documents submitted to the Sponsor will identify the subjects exclusively by number and demographic information. No other personally identifying information should be transmitted to the Sponsor.


Status: Effective 

Sponsor personnel (other than site monitors, lead clinical site manager, person responsible for generating the randomization schedule, and unmasked clinical data managers) involved in reporting, obtaining, and/or reviewing the clinical evaluations will be masked to the identity of the contact lens being administered. This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.

This study is open label with randomized subjects to use either DAILIES TOTAL1 or Acuvue Oasys 1-Day for the duration of the 4-week treatment period.

Visual acuity is the primary endpoint and the study is controlled DAILIES TOTAL1 or Acuvue Oasys 1-Day wearers will be excluded.

### 8.2 Unmasking of the Study Treatment

Not applicable; this study is open-label.

#### 9 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

### 9.1 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the eCRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Study monitors are appointed by the Study Sponsor and are independent of study site staff. If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents should include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)


Status: Effective 

 Records regarding medical histories and the use of concomitant therapies prior to and during the study

• Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the eCRF are consistent with the original source data.

Only designated individuals may complete the eCRFs. The eCRFs will be submitted at regular intervals following the clinical study visit schedule. It is expected that all data reported will have corresponding entries in the source documents. The Principal Investigator is responsible for reviewing and certifying that the eCRFs are accurate and complete. The only subject identifiers recorded on the eCRFs will be subject number, and subject demographic information.

#### 9.2 Data Review and Clarifications

Upon completion of the eCRFs, a targeted review of the eCRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. Additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's eCRFs.

# 9.3 Regulatory Documentation and Records Retention

The Investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the Sponsor and the Investigator's files will be reviewed as part of the ongoing study monitoring. Financial disclosure is not subject to regulatory inspection and should be kept separately.

Additionally, the Investigator must keep study records and source documents until the Sponsor provides written approval for their destruction. If the Investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, the Sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations (generally 2 years after discontinuing clinical development or after the last marketing approval).


Status: Effective 

#### 10 ETHICS AND COMPLIANCE

This trial will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and the referenced directives, regulations, guidelines, and/or standards.

### 10.1 Compliance

The Investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The Investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records.

### 10.2 Institutional Review Board (IRB)

This trial requires IRB approval prior to initiation. This protocol, subject informed consent, and subsequent amendments will be reviewed and approved by an IRB.

Before clinical study initiation, this protocol, the ICF (and assent form, if applicable), any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB. The Investigator must provide documentation of the IRB approval to the Study Sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), ICF, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB must be provided with a copy of the Package Insert, any periodic safety updates, and all other information as required by local regulation and/or the IRB. At the end of the study, the Investigator must notify the IRB about the study's completion. The IRB also must be notified if the study is terminated prematurely. Finally, the Investigator must report to the IRB on the progress of the study at intervals stipulated by the IRB.

Voluntary informed consent must be obtained from every subject (and/or legal representative, as applicable) prior to the initiation of any screening or other study-related procedures. The Investigator must have a defined process for obtaining consent. Specifically, the Investigator, or delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the Investigator, and if required by local regulation, other qualified personnel. The Investigator must provide the subject with


Status: Effective 

a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and Sponsor-designated personnel. The Investigator must keep the original, signed copy of the consent and must provide a duplicate copy to each subject according to local regulations. Following this study, the subject will return to their eye care professional for their routine eye care and contact lenses.

#### 11 PROTOCOL AMENDMENT HISTORY

| Version | Brief Description and Rationale |
|---------|----------------------------------|
| 1 | Initial Version of this document |

#### 12 REFERENCES

### 12.1 References applicable for all clinical trials

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- ISO 14155:2011 Clinical investigation of medical devices for human subjects Good clinical practice

# 12.1.1 US references applicable for clinical trials

- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators
- The California Bill of Rights

#### 12.2 References for this clinical trial

Not applicable.


Status: Effective

| Date/Time<br>(mm/dd/yyyy GMT): | Signed by: | Justification: |
|--------------------------------|------------|------------------------------|
| 07/19/2018 20:04:50 | | Global Device Medical Safety |
| 07/20/2018 09:27:32 | | Clinical Project Lead |
| 07/20/2018 15:20:06 | | biostatistics |